CLINICAL TRIAL: NCT01142193
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of USL255 as Adjunctive Therapy in Patients With Refractory Partial-Onset Seizures
Brief Title: Study to Evaluate the Safety and Effectiveness of USL255 in Patients With Refractory Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P09-004; 2009-016996-31 (EudraCT Number)
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; partial onset seizure; adjunctive therapy
MeSH Terms: conditions — Epilepsy | interventions — Topiramate

ARMS (2):
- USL255 (Experimental)
  Interventions: Drug: USL255
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: USL255
  Arms: USL255
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of USL255 as adjunctive therapy in patients with refractory partial onset-seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of partial-onset seizures with or without secondary generalization for at least 12 months prior to Visit 1.
* Currently on a stable dosing regimen of 1 to 3 AEDs for at least 4-weeks prior to Visit 1 (12 weeks for phenobarbital and primidone).
* Have a minimum of 8 partial-onset seizures and no more than 21 consecutive seizure free days, during the 8-week baseline.

Exclusion Criteria:

* Have a history of seizure episodes lasting less than 30 minutes in which several seizures occur with such frequency that the initiation and completion of each individual seizure cannot be distinguished, within 3 months prior to Visit 1.
* Have a history of pseudoseizures, or status epilepticus, within 3 months prior to Visit 1.
* Have a history of metabolic acidosis, nephrolithiasis, ureterolithiasis, or narrow angle glaucoma.
* Have a history of suicidal attempts, suicidal ideation, or uncontrolled psychiatric illness within 2 years of Visit 1.
* Currently taking, or have taken felbamate within the past 18 months, or have taken vigabatrin in the past.
* Have taken topiramate within the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (19):
  - Phoenix, Arizona
  - Ventura, California
  - Gainesville, Florida
  - Gulf Breeze, Florida
  - Jacksonville, Florida
  - Pensacola, Florida
  - Port Charlotte, Florida
  - Boise, Idaho
  - Lexington, Kentucky
  - Waldorf, Maryland
  - Chesterfield, Missouri
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Toledo, Ohio
  - Dallas, Texas
  - Temple, Texas
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Salta
  - Villa Nueva
- Australia (7):
  - Bedford Park
  - Clayton
  - Fitzory
  - Heidelberg West
  - Parkville
  - Randwick
  - Woodville
- Belgium (3):
  - Bruges
  - Duffel
  - Leuven
- Greenfield Park, Canada
- Chile (2):
  - Santiago
  - Valdivia
- Germany (2):
  - Bonn
  - München
- Greece (2):
  - Athens
  - Thessaloniki
- Budapest, Hungary
- India (5):
  - Bangalore
  - Dehradun
  - Hyderabad
  - Mangalore
  - New Delhi
- Israel (6):
  - Ashkelon
  - Haifa
  - Holon
  - Nahariya
  - Petah Tikva
  - Ramat Gan
- Auckland, New Zealand
- Poland (5):
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Russia (6):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara
  - Tyumen
  - Yaroslavi
- Cape Town, South Africa
- Spain (4):
  - Badalona
  - Barakaldo
  - Granada
  - Madrid

REFERENCES:
- [Derived] Hogan RE, Blatt I, Lawson B, Nagaraddi V, Fakhoury TA, Anders B, Clark AM, Laine D, Halvorsen MB, Chung SS. Efficacy of once-daily extended-release topiramate (USL255): a subgroup analysis based on the level of treatment resistance. Epilepsy Behav. 2014 Dec;41:136-9. doi: 10.1016/j.yebeh.2014.09.061. Epub 2014 Oct 21. PMID 25461205
- [Derived] Chung SS, Fakhoury TA, Hogan RE, Nagaraddi VN, Blatt I, Lawson B, Arnold S, Anders B, Clark AM, Laine D, Meadows RS, Halvorsen MB; PREVAIL Study Group. Once-daily USL255 as adjunctive treatment of partial-onset seizures: randomized phase III study. Epilepsia. 2014 Jul;55(7):1077-87. doi: 10.1111/epi.12660. Epub 2014 Jun 5. PMID 24902983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 16 countries (Argentina, Australia, Belgium, Canada, Chile, Germany, Greece, Hungary, India, Israel, New Zealand, Poland, Russia, South Africa, Spain, and United States). At least 1 subject was enrolled at 66 study centers, of which 60 study centers randomly assigned at least 1 subject to study drug.
Pre-assignment Details: Subject had to have a minimum of 8 partial-onset seizures and no more than 21 consecutive seizure free days during the 8-week baseline to be randomized into the trial.
Groups:
- USL255: Titration of 50 mg in weekly increments over 3 weeks to 200 mg
- Placebo: Placebo
Period: Overall Study
Arm/Group | USL255 | Placebo
Started | 124 | 125
Completed | 103 | 114
Not Completed | 21 | 11
Not completed — Adverse Event | 12 | 4
Not completed — Lack of Efficacy | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Discontinuation Criterion Met | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | USL255 | Placebo | Total
Number analyzed (Participants) | 124 | 125 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (10.97) | 37.6 (11.11) | 37.6 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction From Baseline in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Plus Maintenance Phase Compared to Baseline.
Time Frame: 11 weeks
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Median (Full Range); unit: Percent Reduction
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percent Reduction | 39.5 [-227.3 to 100.0] | 21.65 [-531.2 to 100.0]
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p < .001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 17.85
Statistical Analysis 2: Comparison: USL255 vs Placebo; Test type: Superiority or Other; Hodges-Lehmann; Median Difference (Net) = 18.5, 95% CI 2-sided [8.53 to 28.1]

2. Secondary Outcome: Proportion of Subjects With ≥50% Reduction (Responder Rate) in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Plus Maintenance Phase Compared to Baseline.
Time Frame: 11 weeks
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percentage of participants | 37.9 | 23.2
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p = 0.013, Fisher Exact; Difference in Percentages = 14.7

3. Secondary Outcome: Proportion of Subjects With ≥50% Reduction (Responder Rate) in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Phase Compared to Baseline.
Time Frame: 3 weeks (weeks 1-3)
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percentage of participants | 33.9 | 17.6
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; Analysis was stratified by Geographic Region; Difference in Percentages = 16.3

4. Secondary Outcome: Percent Reductions From Baseline in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Phase Compared to Baseline.
Time Frame: 3 weeks (weeks 1-3)
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Median (Full Range); unit: Percent Reduction
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percent Reduction | 33.93 [-200.00 to 100.0] | 8.57 [-158.3 to 100.0]
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 25.36

5. Secondary Outcome: Percent Reduction From Baseline in Weekly (7 Day) All Seizure Frequency During the Titration Plus Maintenance Phase.
Time Frame: 11 weeks
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Median (Full Range); unit: Percent Reduction
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percent Reduction | 39.50 [-227.3 to 100.0] | 21.65 [-531.2 to 100.0]
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 17.85

6. Secondary Outcome: Proportion of Subjects With ≥25%, ≥75%, and 100% Reduction in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Phases Compared to Baseline.
Time Frame: 3 weeks (weeks 1-3)
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percentage of participants
  ≥25% reduction in seizure rate | 56.5 | 34.4
  ≥75% reduction in seizure rate | 16.9 | 7.2
  100% reduction in seizure rate | 12.1 | 3.2

7. Secondary Outcome: Proportion of Subjects With ≥25%, ≥75%, and 100% Reduction in Weekly (7 Day) Partial-onset Seizure Frequency During the Titration Plus Maintenance Phase Compared to Baseline.
Time Frame: 11 weeks
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 124 | 125
Percentage of participants
  ≥25% reduction in seizure rate | 66.9 | 46.4
  ≥75% reduction in seizure rate | 15.3 | 4.8
  100% reduction in seizure rate | 3.2 | 1.6

8. Secondary Outcome: Proportion of Subjects With ≥25%, ≥75%, and 100% Reduction in Weekly (7 Day) Partial-onset Seizure Frequency During the Maintenance Phase Compared to Baseline.
Time Frame: 8 weeks (weeks 4-11)
Population: Intent-to-treat (ITT): all subjects who were randomized and received at least 1 dose of study drug. Note: Sample size is less than for primary outcome because some subjects discontinued study prior to the maintenance phase.
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 113 | 120
Percentage of participants
  ≥25% reduction in seizure rate | 72.6 | 46.7
  ≥75% reduction in seizure rate | 26.5 | 9.2
  100% reduction in seizure rate | 7.1 | 3.3

9. Secondary Outcome: Percent Reduction From Baseline in Weekly (7 Day) Partial-onset Seizure Frequency During the Maintenance Phase Compared to Baseline.
Time Frame: 8 weeks (weeks 4-11)
Population: as for outcome 8
Measure: Median (Full Range); unit: Percent Reduction
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 113 | 120
Percent Reduction | 45.70 [-237.5 to 100.0] | 22.09 [-747.4 to 100.0]
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 23.61

10. Secondary Outcome: Proportion of Subjects ≥50% Reduction (Responder Rate) in Weekly (7 Day) Partial-onset Seizure Frequency During the Maintenance Phase Compared to Baseline.
Time Frame: 8 weeks (weeks 4-11)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | USL255 | Placebo
Number analyzed (Participants) | 113 | 120
Percentage of participants | 44.2 | 30.8
Statistical Analysis 1: Comparison: USL255 vs Placebo; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel; Analysis was stratified by Geographic Region; Difference in Percentages = 13.4

ADVERSE EVENTS:
Time Frame: Adverse events with onset after the start of study medication and up to 30 days after the last dose of study drug are reported.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE. If a subject experienced more than 1 AE in a system organ class (SOC), the subject is counted only once for that SOC.
Arm/Group | USL255 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/124 | 2/125
Other Adverse Events (participants affected / at risk) | 35/124 | 14/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | USL255 (N=124) | Placebo (N=125)
Lobar Pneumonia (Infections and infestations) | 1 | 0
Physical Assault (Social circumstances) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Epileptic Psychosis (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | USL255 (N=124) | Placebo (N=125)
Somnolence (Nervous system disorders) | 15 | 3
Dizziness (Nervous system disorders) | 9 | 7
Paraesthesia (Nervous system disorders) | 8 | 3
Weight Decreased (Investigations) | 8 | 0
Fatigue (General disorders) | 7 | 6
Headache (Nervous system disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No